CLINICAL TRIAL: NCT02059902
Title: Continuous Lidocaine Infusion for Management of Perioperative Burn Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-105
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Thermal Burns
Keywords: Pain management; Narcotic consumption; Skin graft
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal pain management (Placebo Comparator): Normal saline (bolus followed by continuous infusion)
  Interventions: Other: Placebo
- Lidocaine (Experimental): Lidocaine (Pre-operative = 1.5kg/mg over a minimum of 30 minutes; peri-operative = 2.0mg/kg/hour; Post-operative = 1.5kg/mg/hour)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine infusion runs for a total of 24 hours
  Arms: Lidocaine
Other: Placebo — Normal saline runs for a total of 24 hours
  Arms: Normal pain management

SUMMARY:
Thermal injury results in one of the most intense and prolonged forms of pain the body can experience. Opioid narcotics are the most powerful drugs for acute and chronic pain, and their use in the perioperative period has been the mainstay of treatment; although medication requirements in burn patients are often underestimated. More medication may not be the answer, as relatively large doses of short acting opioids in the operative theater are associated with greater postoperative opioid consumption and higher pain scores. Furthermore, extensive use of opioids has resulted in the development of by hyperalgesia and allodynia. Lidocaine is an amide local anesthetic that has analgesic, anti-hyperalgesic, antiarrhythmic, and anti-inflammatory properties. Over the past 25 years, systemic lidocaine has been used for perioperative pain management in a variety of surgical procedures. The design of this study will examine if lidocaine will reduce the pain scores and narcotic utilization in patients undergoing surgical procedures for burn injuries. The intervention group will receive a bolus dose of lidocaine followed by a continuous infusion over 24 hours. The control group will get an equal volume of saline. The investigators will compare pain scores, opioid use, and narcotic equivalents based on body weight and burn surface area (BSA) grafted.

ELIGIBILITY:
Inclusion Criteria:

* Burn patient ≥ 18 years of age
* Burn patient scheduled to go to OR for excision and/or grafting procedure

Exclusion Criteria:

* Burn patient < 18 years of age
* Intubated patient on sedation drip
* Prolonged hypotension defined as Systolic Blood Pressure (SBP) < 90 mm/Hg for greater than 30 minutes in the pre-op area
* Severe underlying cardiovascular disease (documented ejection fraction < 40%)
* Documented conduction block, bradycardia or active congestive heart failure
* Documented active gastritis or ulcers
* Previous steroid medication history if documented adrenal insufficiency
* Patient with documented liver disease
* Patient with epilepsy or known seizure disorder
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Mohr, MD, Principal Investigator — Regions Hospital; Sandi Wewerka, MPH, Study Director — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 patients were consented during the study period, 28 patients randomized and treated: 14 placebo vs. 14 lidocaine. Patients were excluded after signing consent for: arriving to the pre-op area wearing a Lidocaine patch, changes in surgery times, lack of grafting/surgery needs, and medical contraindications (such as lidocaine with metoprolol).
Period: Overall Study
Arm/Group | Normal Pain Management | Lidocaine
Started | 18 | 18
Completed | 14 | 14
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Pain Management | Lidocaine | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Full Range); unit: years] | 43.5 [29 to 69] | 35.7 [19 to 58] | 39.48 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Total Burn Surface Area [Mean (Full Range); unit: total percentage of body area burned] | 17.77 [1 to 68] | 11.18 [1 to 48.39] | 14.48 [1 to 68]

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Consumption (Measured in mg/kg Narcotic Consumption)
Description: The infusion was initiated at 1.5mg/kg for 30 minutes prior to surgery start, followed by a 2.0 mg/kg/hr infusion at the time of incision start. The rate was reduced to 1.5mg/kg/hr for the remainder of the 24 hour period. A standardized post-operative pain management strategy (morphine and oxycodone) was followed by clinical staff, based on a standardized pain scale rating tool. The difference in narcotic consumption and number of pain medication doses over the 72-hour post-operative period was compared using an unadjusted Wilcoxon rank sum test due to non-normal data distribution.
Time Frame: 24-hours post surgery
Measure: Median (Inter-Quartile Range); unit: mg/kg narcotic consumption
Arm/Group | Normal Pain Management | Lidocaine
Number analyzed (Participants) | 14 | 14
mg/kg narcotic consumption | 57.5 [35 to 105] | 67.75 [50 to 134]

ADVERSE EVENTS:
Arm/Group | Normal Pain Management | Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes